CLINICAL TRIAL: NCT03648021
Title: NEUROTHERM: The Effect of Paracetamol on Brain Temperature in Acute Brain Injury in a Neuro Critical Care Unit: A Randomized Controlled Trial
Brief Title: The Effect of Paracetamol on Brain Temperature
Acronym: NEUROTHERM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDY_2017_19
Record Dates: First submitted 2018-08-03; First posted 2018-08-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paracetamol (acetaminophen) (Active Comparator): patient will receive1 gramme of paracetamol intravenously
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): patient will receive 100 ml of chlorure de sodium 0,9% intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — >50kg: Paracetamol 1 gramme in a solution of 10mg/mL administred intravenously. 1 dose
  >50kg: Paracetamol 15mg/kg/dose in a solution 10mg/mL administred intravenously. 1 dose
  Other Names: acetaminophen
  Arms: paracetamol (acetaminophen)
Drug: Placebo — 100mL of chlorure de sodium 0.9% administred intravenously. 1 dose
  Arms: Placebo

SUMMARY:
The main objective of this study is to compare the effect of intravenous paracetamol administration on mean brain temperature (measured between H0 and H6) in patients with cerebral hyperthermia versus placebo.

The investigators will measure brain temperature using a thermistor that will be connected to the intracranial pressure transducer.

ELIGIBILITY:
Inclusion Criteria

* 18-year or older patients
* Patient hospitalized in neuro-critical care for:
* Arachnoid hemorrhage
* Intra parenchymatous hematoma
* stroke
* Acute brain Severe injury
* Post-operative complication of an act of neurosurgery or programmed neuroradiology
* Sedation and mechanical ventilation planned > 2 days
* Monitoring of intracranial temperature and pressure by intraparenchymal sensor (Sophysa®)
* Brain temperature > 38.5°C for more than 30 minutes

Exclusion Criteria

* Known hypersensitivity to paracetamol or mannitol (excipient with known effect)
* Severe hepatocellular insufficiency (ASAT or ALAT > 5N, or bilirubin > 2N)
* Pharmacological intervention (administration of corticosteroids, NSAIDs or paracetamol) or physical intervention (external cooling technique) that may influence temperature in the last 6 hours.
* Pregnant or breastfeeding women
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Comparison of mean brain temperature measured between H0 and H6 following administration of treatment between the two groups (the group treated with paracetamol and the placebo group) | Six hours after administration of treatment
  measurement of intracerebral temperature in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Marine de Mesmay, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] de Mesmay M, Geral L, Gregoire C, Roy M, Welschbillig S, Le Cossec C, Engrand N. Effect of Paracetamol on Cerebral Temperature in Febrile Brain-Injured Patients. The NEUROTHERM Study: A Randomized Controlled Pharmacodynamic Trial. Crit Care Med. 2026 Jan 1;54(1):108-118. doi: 10.1097/CCM.0000000000006951. Epub 2025 Nov 11. PMID 41217349